CLINICAL TRIAL: NCT03040167
Title: The Pectoral Block for Breast Augmentation Surgery: a Volunteers' and Patients' Study.
Brief Title: The Pectoral Block for Breast Augmentation Surgery
Acronym: BPCAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pierre Beaulieu (Other)
Collaborators: Ministere de la Sante et des Services Sociaux (Other)
Responsible Party: Sponsor-Investigator, Pierre Beaulieu, Professor of anesthesiology, Centre hospitalier de l'Université de Montréal (CHUM)
Organization: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17.091
Record Dates: First submitted 2017-01-29; First posted 2017-02-02 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2018-03

CONDITIONS: Pain, Postoperative; Anesthesia; Regional
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): PEC 1 block with injection of 0.4 mL/kg of normal saline under echoguidance.
  Interventions: Procedure: PEC 1 block; Drug: Normal saline
- Treatment group (Active Comparator): PEC 1 block with injection of 0.4 mL/kg of 0.25% bupivacaine with 1/400 000 epinephrine under echoguidance.
  Interventions: Procedure: PEC 1 block; Drug: Bupivacaine with epinephrine

INTERVENTIONS:
Procedure: PEC 1 block — Under echoguidance, injection of the substance of interest between the major and minor pectoral muscles.
  Other Names: pectoral block; pecblock
Drug: Bupivacaine with epinephrine — Treatment group
  Arms: Treatment group
Drug: Normal saline — Placebo group
  Arms: Control group

SUMMARY:
The pectoral block is a recently developed regional anesthetic technique that can be used for the treatment of postoperative pain after breast surgery. Injection of local anesthetic between the major and the minor pectoral muscles is defined as the pectoral (PEC) 1 block. This block has not been well characterized in terms of its blocking effects on motor and sensitive nerves (medial and lateral pectoral nerves and intercostal nerves). This clinical trial is divided into two sections: a volunteer study and a patient study.

For the volunteer study, the aim is to assess the sensory territory affected by injection of local anesthetics through a PEC 1 block and to assess motor function in terms of strength of adduction of the affected limb using a dynamometer.

In a prospective, randomized, controlled and double blind study, the aim is to assess the postoperative pain relieving properties of the PEC 1 block in patients undergoing bilateral breast augmentation surgery.

ELIGIBILITY:
Inclusion Criteria:

* breast augmentation surgery
* registration at régie d'assurance maladie du Québec (RAMQ) (social services)

Exclusion Criteria:

* known bleeding disorder
* anticoagulant intake
* infection at site of PEC 1 block
* pregnant or breast-feeding women
* allergy to bupivacaine
* chronic pain including fibromyalgia with regular analgesic consumption
* under recreational drugs or alcohol at doses above canadian recommendations
* muscle relaxants intake
* patients already operated for breast augmentation or mastectomy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score at rest | Within the first 10 min after arrival to the postanesthesia care unit (PACU)
  Pain score using a verbal numerical scale (0-10) in one breast (bupivacaine) compared to the other breast (placebo)

SECONDARY OUTCOMES:
Postoperative pain score on movement | Within the first 10 min after arrival to the postanesthesia care unit (PACU)
  Pain score using a verbal numerical scale (0-10) in one breast (bupivacaine) compared to the other breast (placebo)
Postoperative pain score at rest | 15 min, 30 min, 60 min, 12h and 24 h after time of arrival in the PACU and immediately after discharge from PACU
  Pain score using a verbal numerical scale (0-10) in one breast (bupivacaine) compared to the other breast (placebo)
Incidence of nausea and/or vomiting | 15 min, 30 min, 60 min, 12h and 24 h after time of arrival in the PACU and immediately after discharge from PACU
  Presence or absence of nausea and/or vomiting
Surgical bleeding | After surgery for 24 hours
  Presence or not of surgical bleeding from wounds, drains eventually leading to surgical exploration
Hematoma | After surgery for 24 hours
  Presence or absence of hematoma at PEC 1 block injection
Postoperative well-being | At 24 hours after surgery
  Analgesic intake

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - CHUM, Montreal, Quebec
  - CISSS des Laurentides, Saint-Jérôme, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Desroches J, Belliveau M, Bilodeau C, Landry M, Roy M, Beaulieu P. Pectoral nerves I block is associated with a significant motor blockade with no dermatomal sensory changes: a prospective volunteer randomized-controlled double-blind study. Can J Anaesth. 2018 Jul;65(7):806-812. doi: 10.1007/s12630-018-1122-2. Epub 2018 Mar 29. PMID 29600482